CLINICAL TRIAL: NCT03569098
Title: A Multiple-dose, Double-blind, Randomised, Placebo-controlled Study to Evaluate the Efficacy and Safety of Dysport for the Treatment of Pain Associated With Hallux Abducto Valgus
Brief Title: Dysport in Hallux Abducto Valgus (HAV) Phase IIa
Acronym: DYSTANCE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D-FR-52120-237
Record Dates: First submitted 2018-06-14; First posted 2018-06-26 (Actual); Results first posted 2021-07-02 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-07

CONDITIONS: Hallux Abducto Valgus
MeSH Terms: interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dysport Dose 1 (Experimental): Intramuscular injection of Dysport on day 1 of double-blind period, followed by up to 2 open-label injections during open-label cycles, during approximately 36 weeks.
  Interventions: Biological: Botulinum toxin type A
- Dysport Dose 2 (Experimental): Intramuscular injection of Dysport on day 1 of double-blind period, followed by up to 2 open-label injections during open-label cycles, during approximately 36 weeks.
  Interventions: Biological: Botulinum toxin type A
- Placebo (Placebo Comparator): Intramuscular injection of Placebo on day 1 of cycle 1 (double-blind period)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Botulinum toxin type A — Investigators will inject the reconstituted solution into foot muscles.
  Other Names: AbobotulinumtoxinA (Dysport®); Clostridium botulinum toxin type A haemagglutinin complex (BTX-A-HAC)
  Arms: Dysport Dose 1; Dysport Dose 2
Drug: Placebo — Investigators will inject the reconstituted solution into foot muscles.
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of treatment with multiple doses of Dysport in adults suffering from clinically significant pain associated with HAV who have not undergone surgery for their condition.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of HAV
* Painful HAV in the study foot at Baseline

Exclusion Criteria:

* Flat or square metatarsal head, metatarsus primus elevates, or severe cavus/planus in the study foot
* Other podiatric or orthopedic condition which would interfere with the evaluation of pain and/or function
* Medical history or clinical evidence of any vascular disease and/or diabetic condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2020-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (29):
- United States (29):
  - NEA Baptist Clinic, Jonesboro, Arkansas
  - Applied Research Center of Arkansas, Inc, Little Rock, Arkansas
  - Center for Clinical Research Inc., Castro Valley, California
  - Limb Preservation Platform, Inc., Fresno, California
  - Southwestern Academic Limb Salvage Alliance, Los Angeles, California
  - Foot and Ankle Clinic, Los Angeles, California
  - University Foot and Ankle Institute, Santa Monica, California
  - Center for Spine and Orthopedics, Thornton, Colorado
  - LCC Medical Research Institute, Miami, Florida
  - Conquest Research, Orlando, Florida
  - Doctors Research Network, South Miami, Florida
  - Clinical Research, West Palm Beach, Florida
  - Podiatry 1st, Belleville, Illinois
  - Weil Foot & Ankle Institute, Des Plaines, Illinois
  - Rosalind Franklin Clinic, North Chicago, Illinois
  - Foot and Ankle Center of Illinois, Springfield, Illinois
  - The Chesapeake Research Group, Pasadena, Maryland
  - Dr. Allen M. Jacobs and Associates, St Louis, Missouri
  - Ankle and Foot Care Centers, Youngstown, Ohio
  - Medical Research International, Oklahoma City, Oklahoma
  - Foot and Ankle Center, Bryn Mawr, Pennsylvania
  - Harrisburg Foot and Ankle Center, INC, Harrisburg, Pennsylvania
  - Futuro Clinical Trials, LLC, McAllen, Texas
  - Bio X Cell Research, San Antonio, Texas
  - Texas Gulf Coast Medical Group, Webster, Texas
  - Summit Foot & Ankle, Salt Lake City, Utah
  - Harrisonburg Foot and Ankle Clinic, Harrisonburg, Virginia
  - 1Foot 2Foot Centre for Foot and Ankle Care, PC, Suffolk, Virginia
  - Martinsville Research Institute, Inc., Salem, West Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase II double-blind study was conducted at 27 sites in the United States between 19 June 2018 and 22 May 2020 in adult participants suffering from clinically significant hallux abducto valgus (HV) who have not undergone surgery for their condition.
Pre-assignment Details: The study consisted of a screening period (up to 3 weeks), followed by a double-blind treatment period (Cycle 1). From Week 12, retreatment criteria were evaluated every 4 weeks to determine eligibility to receive treatment in the open-label period (Cycles 2 and 3). Total study duration was a maximum of 36 weeks. A total of 186 participants were randomized in a 1:1:1 ratio to 1 of 3 treatment groups (placebo, Dysport 300 units (U) and Dysport 500 U) in the double-blind treatment period.
Groups:
- Placebo: On Cycle 1 Day 1 in the double-blind treatment period, participants received a single dose of placebo (matching with Dysport) intramuscular injection distributed between 4 injection points in the 4 targeted muscles of the study foot.
  Following the double-blind treatment period, all participants who met retreatment criteria were treated during the open-label period with Dysport 300 U on Cycle 2 Day 1 and either Dysport 300 U or 500 U on Cycle 3 Day 1.
  The 4 targeted muscles of the study foot were the oblique head of the adductor hallucis muscle, the transverse head of the adductor hallucis muscle, the flexor hallucis brevis muscle and the extensor hallucis brevis muscle.
- Dysport 300 U: On Cycle 1 Day 1 in the double-blind treatment period, participants received a single dose of Dysport 300 U intramuscular injection distributed between 4 injection points (75 U each) in the 4 targeted muscles of the study foot.
  Following the double-blind treatment period, all participants who met retreatment criteria were treated during the open-label period with Dysport 300 U on Cycle 2 Day 1 and either Dysport 300 U or 500 U on Cycle 3 Day 1.
  The 4 targeted muscles of the study foot were the oblique head of the adductor hallucis muscle, the transverse head of the adductor hallucis muscle, the flexor hallucis brevis muscle and the extensor hallucis brevis muscle.
- Dysport 500 U: On Cycle 1 Day 1 in the double-blind treatment period, participants received a single dose of Dysport 500 U intramuscular injection distributed between 4 injection points (125 U each) in the 4 targeted muscles of the study foot.
  Following the double-blind treatment period, all participants who met retreatment criteria were treated during the open-label period with Dysport 300 U on Cycle 2 Day 1 and either Dysport 300 U or 500 U on Cycle 3 Day 1.
  The 4 targeted muscles of the study foot were the oblique head of the adductor hallucis muscle, the transverse head of the adductor hallucis muscle, the flexor hallucis brevis muscle and the extensor hallucis brevis muscle.
Period: Double-Blind Treatment Cycle 1
Arm/Group | Placebo | Dysport 300 U | Dysport 500 U
Started | 63 | 63 | 60
Received Study Medication | 61 | 63 | 56
Completed (Completed the double-blind treatment cycle 1.) | 55 | 53 | 49
Not Completed | 8 | 10 | 11
Not completed — Withdrawal by Subject | 5 | 2 | 5
Not completed — Study terminated by sponsor | 0 | 6 | 3
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Technical problems | 0 | 0 | 2
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Protocol deviation | 0 | 1 | 0
Not completed — Other | 1 | 0 | 1
Period: Open-Label Treatment Cycle 2
Arm/Group | Placebo | Dysport 300 U | Dysport 500 U
Started | 0 (No participants were treated with placebo during the open-label treatment cycle 2.) | 146 (All participants who met retreatment criteria were treated with Dysport 300 U during the open-label treatment cycle 2.) | 0 (No participants were treated with Dysport 500 U during the open-label treatment cycle 2.)
Completed (Completed the open-label treatment cycle 2.) | 0 | 111 | 0
Not Completed | 0 | 35 | 0
Not completed — Study terminated by sponsor | 0 | 21 | 0
Not completed — Withdrawal by Subject | 0 | 11 | 0
Not completed — Lost to Follow-up | 0 | 3 | 0
Period: Open-Label Treatment Cycle 3
Arm/Group | Placebo | Dysport 300 U | Dysport 500 U
Started | 0 | 8 (Participants were treated with Dysport 300 U during open-label treatment cycle 3 based on investigator judgment following clinical evaluation of the participant at the time of retreatment.) | 56 (Participants were treated with Dysport 500 U during open-label treatment cycle 3 based on investigator judgment following clinical evaluation of the participant at the time of retreatment.)
Completed (Completed the open-label treatment cycle 3.) | 0 | 7 | 50
Not Completed | 0 | 1 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 4
Not completed — Study terminated by sponsor | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Intention-to-Treat (ITT) analysis set included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dysport 300 U | Dysport 500 U | Total
Number analyzed (Participants) | 63 | 63 | 60 | 186
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.3 (13.18) | 48.4 (14.04) | 48.0 (12.24) | 48.2 (13.12)
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 56 | 58 | 57 | 171
  >=65 and <85 years | 7 | 5 | 3 | 15
  >=85 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 60 | 56 | 171
  Male | 8 | 3 | 4 | 15
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 5 | 6 | 12
  Black or African American | 10 | 4 | 9 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  White | 49 | 54 | 43 | 146
  Other | 3 | 0 | 2 | 5
  Hispanic or Latino | 16 | 10 | 16 | 42
  Not Hispanic or Latino | 47 | 53 | 44 | 144

OUTCOME MEASURES:

1. Primary Outcome: Least Square (LS) Mean Change From Baseline in the Daily Numeric Pain Rating Scale (NPRS) Score at Week 8
Description: The NPRS is a widely used and validated unidimensional measure of pain intensity in adults. Participants were asked to rate the intensity of their foot pain during physical activity (example, walking, standing or running) based on an 11-point scale ranging from 0 to 10, where 0 represents "no pain" and 10 represents "worst possible pain". Higher scores indicate a worse outcome. Daily pain intensities were recorded by the participant using an electronic diary (eDiary) for 7 consecutive days prior to each study visit. Baseline was defined as the daily NPRS score averaged over the 7 consecutive days prior to the Baseline visit (Day 1).
Time Frame: Baseline and Week 8 in the double-blind treatment period
Population: The ITT analysis set included all randomized participants. For participants without any available post-Baseline NPRS average scores, the Week 8 average pain score was imputed.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Dysport 300 U | Dysport 500 U
Number analyzed (Participants) | 63 | 63 | 60
units on a scale | -2.04 [-2.66 to -1.41] | -1.71 [-2.33 to -1.10] | -2.40 [-3.03 to -1.77]
Statistical Analysis 1: Comparison: Placebo vs Dysport 300 U; Dysport 300 U versus Placebo; Test type: Superiority; p = 0.7669, Mixed Model for Repeated Measures (MMRM) — One-sided P-value. The model includes the fixed categorical effects of treatment group, visit, treatment group-by-visit interaction, and the stratification factor as fixed categorical covariates and the Baseline value as a fixed continuous covariate; Difference in LS mean = 0.32, 95% CI 2-sided [-0.55 to 1.19], Standard Error of Mean 0.441
Statistical Analysis 2: Comparison: Placebo vs Dysport 500 U; Dysport 500 U versus Placebo; Test type: Superiority; p = 0.2085, MMRM — [p-value comment as in outcome 1, analysis 1]; Difference in LS mean = -0.36, 95% CI 2-sided [-1.24 to 0.51], Standard Error of Mean 0.444

2. Secondary Outcome: LS Mean Change From Baseline in the Daily NPRS Score at Weeks 4 and 12
Description: The NPRS is a widely used and validated unidimensional measure of pain intensity in adults. Participants were asked to rate the intensity of their foot pain during physical activity (example, walking, standing or running) based on an 11-point scale ranging from 0 to 10, where 0 represents "no pain" and 10 represents "worst possible pain". Higher scores indicate a worse outcome. Daily pain intensities were recorded by the participant using an eDiary for 7 consecutive days prior to each study visit. Baseline was defined as the daily NPRS score averaged over the 7 consecutive days prior to the Baseline visit (Day 1).
Time Frame: Baseline and Weeks 4 and 12 in the double-blind treatment period
Population: The ITT analysis set included all randomized participants. For participants without any available post-Baseline NPRS average scores, the Weeks 4 and 12 average pain scores were imputed.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Dysport 300 U | Dysport 500 U
Number analyzed (Participants) | 63 | 63 | 60
units on a scale
  Week 4 | -1.68 [-2.26 to -1.11] | -1.36 [-1.94 to -0.78] | -1.85 [-2.45 to -1.25]
  Week 12 | -1.72 [-2.35 to -1.09] | -1.61 [-2.23 to -1.00] | -2.42 [-3.06 to -1.78]

3. Secondary Outcome: LS Mean Change From Baseline in the Daily Modified Foot Function Index (mFFI) Disability Subscale Score at Weeks 4, 8 and 12
Description: The foot function index (FFI) was developed to assess foot-related pain, disability and activity limitations and later revised to include foot-related health and quality of life. A modified version of FFI specific to this study was used. The mFFI consists of a total of 21 items grouped into 3 subscales: pain (7 questions), disability (9 questions) and activity limitation (5 questions). The mFFI disability subscale is rated using numeric rating scale ranging from 0 to 10, where 0 represents "no difficulty" and 10 represents "so difficult unable to do". For each item, the participant was asked to record the number value which best corresponded to effect of the foot complaints. To obtain a subscale score, the item scores for a given subscale (i.e., pain, disability or activity limitation subscales) were totaled and divided by maximum total possible and then multiplied by 100. Each subscale score, as well as the total score, ranged from 0 to 100. Higher scores indicate a worse outcome.
Time Frame: Baseline and Weeks 4, 8 and 12 in the double-blind treatment period
Population: The ITT analysis set included all randomized participants. The results are presented for the participants with data available at Baseline and specific time points.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Dysport 300 U | Dysport 500 U
Number analyzed (Participants) | 52 | 53 | 47
units on a scale
  Week 4: number analyzed (Participants) | 52 | 50 | 46
  Week 4 | -17.95 [-23.06 to -12.84] | -15.29 [-20.47 to -10.12] | -16.87 [-22.27 to -11.48]
  Week 8: number analyzed (Participants) | 49 | 52 | 47
  Week 8 | -22.44 [-28.00 to -16.87] | -18.68 [-24.19 to -13.17] | -21.26 [-27.05 to -15.48]
  Week 12: number analyzed (Participants) | 48 | 53 | 46
  Week 12 | -17.21 [-23.11 to -11.31] | -21.04 [-26.80 to -15.27] | -21.50 [-27.61 to -15.39]

4. Secondary Outcome: LS Mean Change From Baseline in the Daily mFFI Pain Subscale Score at Weeks 4, 8 and 12
Description: The FFI was developed to assess foot-related pain, disability and activity limitations and later revised to include foot-related health and quality of life. A modified version of the FFI specific to this study was used. The mFFI consists of a total of 21 items grouped into 3 subscales: pain (7 questions), disability (9 questions) and activity limitation (5 questions). The mFFI pain subscale is rated using numeric rating scale ranging from 0 to 10, where 0 represents "no pain" and 10 represents "worst pain imaginable". For each item, the participant was asked to record the number value which best corresponded to the effect of the foot complaints. To obtain a subscale score, the item scores for a given subscale (i.e., pain, disability or activity limitation subscales) were totaled and divided by the maximum total possible and then multiplied by 100. Each subscale score, as well as the total score, ranged from 0 to 100. Higher scores indicate a worse outcome.
Time Frame: Baseline and Weeks 4, 8 and 12 in the double-blind treatment period
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Dysport 300 U | Dysport 500 U
Number analyzed (Participants) | 52 | 53 | 48
units on a scale
  Week 4: number analyzed (Participants) | 52 | 50 | 46
  Week 4 | -17.97 [-23.23 to -12.70] | -15.67 [-21.00 to -10.33] | -19.30 [-24.86 to -13.73]
  Week 8: number analyzed (Participants) | 49 | 52 | 48
  Week 8 | -22.30 [-28.15 to -16.45] | -20.69 [-26.50 to -14.88] | -24.58 [-30.67 to -18.49]
  Week 12: number analyzed (Participants) | 48 | 53 | 46
  Week 12 | -18.94 [-25.05 to -12.83] | -21.74 [-27.72 to -15.76] | -24.30 [-30.64 to -17.96]

5. Secondary Outcome: LS Mean Change From Baseline in the Daily mFFI Total Score at Weeks 4, 8 and 12
Description: The FFI was developed to assess foot-related pain, disability and activity limitations and later revised to include foot-related health and quality of life. A modified version of the FFI specific to this study was used. The mFFI consists of a total of 21 items grouped into three subscales: pain (7 questions), disability (9 questions) and activity limitation (5 questions). The mFFI items are rated using numeric rating scales ranging from 0 to 10, where 0 represents "no pain/no difficulty/none of the time" and 10 represents "worst pain imaginable/so difficult unable to do/all of the time" for pain, disability and activity limitation subscales, respectively. For each item, the participant was asked to record the number value which best corresponded to the effect of the foot complaints. To obtain a total score, the scores of all 3 subscales were totaled and divided by 3. Each subscale score, as well as the total score, ranged from 0 to 100. Higher scores indicate a worse outcome.
Time Frame: Baseline and Weeks 4, 8 and 12 in the double-blind treatment period
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Dysport 300 U | Dysport 500 U
Number analyzed (Participants) | 52 | 53 | 47
units on a scale
  Week 4: number analyzed (Participants) | 52 | 50 | 46
  Week 4 | -14.87 [-18.98 to -10.75] | -12.80 [-16.96 to -8.64] | -15.10 [-19.45 to -10.76]
  Week 8: number analyzed (Participants) | 49 | 52 | 47
  Week 8 | -18.82 [-23.32 to -14.32] | -16.16 [-20.62 to -11.69] | -18.79 [-23.48 to -14.11]
  Week 12: number analyzed (Participants) | 48 | 53 | 46
  Week 12 | -15.65 [-20.48 to -10.82] | -17.45 [-22.18 to -12.72] | -18.89 [-23.90 to -13.88]

6. Secondary Outcome: LS Mean Change From Baseline in the Daily mFFI Activity Limitation Subscale Score at Weeks 4, 8 and 12
Description: The FFI was developed to assess foot-related pain, disability and activity limitations and later revised to include foot-related health and quality of life. A modified version of the FFI specific to this study was used. The mFFI consists of a total of 21 items grouped into 3 subscales: pain (7 questions), disability (9 questions) and activity limitation (5 questions). The mFFI activity limitation subscale is rated using numeric rating scale ranging from 0 to 10, where 0 represents "none of the time" and 10 represents "all of the time". For each item, the participant was asked to record the number value which best corresponded to the effect of the foot complaints. To obtain a subscale score, the item scores for a given subscale (i.e., pain, disability or activity limitation subscales) were totaled and divided by the maximum total possible and then multiplied by 100. Each subscale score, as well as the total score, ranged from 0 to 100. Higher scores indicate a worse outcome.
Time Frame: Baseline and Weeks 4, 8 and 12 in the double-blind treatment period
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Dysport 300 U | Dysport 500 U
Number analyzed (Participants) | 52 | 53 | 48
units on a scale
  Week 4: number analyzed (Participants) | 52 | 50 | 46
  Week 4 | -9.02 [-12.08 to -5.96] | -7.00 [-10.08 to -3.91] | -9.03 [-12.28 to -5.79]
  Week 8: number analyzed (Participants) | 49 | 52 | 48
  Week 8 | -12.12 [-15.52 to -8.71] | -8.81 [-12.17 to -5.45] | -10.62 [-14.17 to -7.07]
  Week 12: number analyzed (Participants) | 48 | 53 | 46
  Week 12 | -11.09 [-14.79 to -7.40] | -9.25 [-12.87 to -5.63] | -10.84 [-14.69 to -6.99]

7. Secondary Outcome: LS Mean Change From Baseline in HV Angle at Weeks 4, 8 and 12
Description: The HV angle was measured directly on weight-bearing anteriorposterior radiographs, in which the X-ray beam was angled 15° towards the heel centered on the second tarsometatarsal joint with a source to image-receptor distance of 100 centimeters (cm).
Time Frame: Baseline and Weeks 4, 8 and 12 in the double-blind treatment period
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: degrees
Arm/Group | Placebo | Dysport 300 U | Dysport 500 U
Number analyzed (Participants) | 59 | 62 | 54
degrees
  Week 4 | -0.31 [-1.06 to 0.45] | -0.25 [-0.99 to 0.49] | -0.92 [-1.71 to -0.13]
  Week 8: number analyzed (Participants) | 57 | 59 | 54
  Week 8 | -0.43 [-1.17 to 0.30] | -0.67 [-1.40 to 0.05] | -0.80 [-1.57 to -0.04]
  Week 12: number analyzed (Participants) | 56 | 59 | 51
  Week 12 | 0.30 [-0.44 to 1.05] | -0.68 [-1.41 to 0.04] | -0.45 [-1.22 to 0.33]

8. Secondary Outcome: LS Mean Change From Baseline in Intermetatarsal Angle at Weeks 4, 8 and 12
Description: The intermetatarsal angle was measured directly on weight-bearing anteriorposterior radiographs, in which the X-ray beam was angled 15° towards the heel centered on the second tarsometatarsal joint with a source to image-receptor distance of 100 cm.
Time Frame: Baseline and Weeks 4, 8 and 12 in the double-blind treatment period
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: degrees
Arm/Group | Placebo | Dysport 300 U | Dysport 500 U
Number analyzed (Participants) | 59 | 62 | 54
degrees
  Week 4 | 0.06 [-0.34 to 0.46] | 0.40 [0.01 to 0.79] | 0.16 [-0.25 to 0.58]
  Week 8: number analyzed (Participants) | 57 | 59 | 54
  Week 8 | -0.02 [-0.41 to 0.36] | 0.49 [0.11 to 0.87] | 0.45 [0.05 to 0.85]
  Week 12: number analyzed (Participants) | 56 | 59 | 51
  Week 12 | 0.42 [0.01 to 0.83] | 0.19 [-0.21 to 0.59] | 0.04 [-0.38 to 0.47]

9. Secondary Outcome: Median Time to Retreatment
Description: Time to retreatment was calculated as ([Date of retreatment - previous injection date] + 1) / 7 (week). Time to retreatment was calculated for each cycle and the data presented here for the double-blind treatment period.
Time Frame: Up to 24 weeks in the double-blind treatment period
Population: The safety population included all participants who received at least one dose of study drug administration (including only partial administration). Participants who were not retreated were considered censored at the date of their last visit and not included in the summary but included in the analysis.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo | Dysport 300 U | Dysport 500 U
Number analyzed (Participants) | 61 | 63 | 56
weeks | 12.6 [12 to 13] | 13.1 [13 to 16] | 13.1 [13 to 15]

10. Secondary Outcome: LS Mean Change From Baseline in Patient Global Impression of Severity (PGI-S) of Foot Pain Score at Weeks 4, 8 and 12
Description: An assessment of PGI-S of foot pain was conducted by the participant using a 4-point Likert scale ranging from 0= no pain to 3= severe pain. Higher scores indicate a worse outcome. The PGI-S was assessed by the participant by answering the following question: "How severe was your foot pain while performing physical activities (example, standing, walking or running) over the past week?" (0=no pain; 1=mild pain; 2=moderate pain; 3=severe pain).
Time Frame: Baseline and Weeks 4, 8 and 12 in the double-blind treatment period
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Dysport 300 U | Dysport 500 U
Number analyzed (Participants) | 50 | 53 | 46
units on a scale
  Week 4: number analyzed (Participants) | 50 | 49 | 42
  Week 4 | -0.76 [-0.99 to -0.54] | -0.56 [-0.80 to -0.32] | -0.46 [-0.71 to -0.22]
  Week 8: number analyzed (Participants) | 45 | 47 | 46
  Week 8 | -0.74 [-0.97 to -0.51] | -0.64 [-0.88 to -0.39] | -0.79 [-1.03 to -0.56]
  Week 12: number analyzed (Participants) | 47 | 53 | 41
  Week 12 | -0.58 [-0.82 to -0.35] | -0.59 [-0.82 to -0.36] | -0.60 [-0.85 to -0.35]

11. Secondary Outcome: LS Mean Change From Baseline in PGI-S of Disability Score at Weeks 4, 8 and 12
Description: An assessment of PGI-S of disability was conducted by the participant using a 4-point Likert scale ranging from 0= no disability to 3= severe disability. Higher scores indicate a worse outcome. The PGI-S was assessed by the participant by answering the following question: "How severe was your disability while performing physical activities (example, standing, walking or running) over the past week?" (0=no disability; 1=mild disability; 2=moderate disability; 3=severe disability).
Time Frame: Baseline and Weeks 4, 8 and 12 in the double-blind treatment period
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Dysport 300 U | Dysport 500 U
Number analyzed (Participants) | 50 | 53 | 46
units on a scale
  Week 4: number analyzed (Participants) | 50 | 49 | 41
  Week 4 | -0.47 [-0.70 to -0.25] | -0.57 [-0.82 to -0.32] | -0.42 [-0.68 to -0.16]
  Week 8: number analyzed (Participants) | 45 | 47 | 46
  Week 8 | -0.54 [-0.80 to -0.28] | -0.66 [-0.93 to -0.38] | -0.68 [-0.94 to -0.42]
  Week 12: number analyzed (Participants) | 47 | 53 | 41
  Week 12 | -0.55 [-0.80 to -0.31] | -0.63 [-0.87 to -0.38] | -0.67 [-0.93 to -0.40]

12. Secondary Outcome: LS Mean Patient Global Impression of Improvement (PGI-I) of Foot Pain Score at Weeks 4, 8 and 12
Description: An assessment of PGI-I of foot pain was conducted by the participant using a 7-point Likert scale ranging from -3= very much worse to +3= very much improved. Higher scores indicate a better outcome. The PGI-I was assessed by the participant answering the following question: "Compared to your foot pain prior to the study treatment initiation, your foot pain while performing physical activities (example, standing, walking or running) now is: +3=very much improved; +2=much improved; +1=minimally improved; 0=no change; -1=minimally worse; -2=much worse; -3=very much worse".
Time Frame: Weeks 4, 8 and 12 in the double-blind treatment period
Population: The ITT analysis set included all randomized participants. The results are presented for the participants with data available at specific time points.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Dysport 300 U | Dysport 500 U
Number analyzed (Participants) | 51 | 53 | 46
units on a scale
  Week 4: number analyzed (Participants) | 51 | 50 | 42
  Week 4 | 1.32 [0.98 to 1.65] | 1.32 [0.98 to 1.66] | 1.53 [1.17 to 1.90]
  Week 8: number analyzed (Participants) | 45 | 47 | 46
  Week 8 | 1.30 [0.94 to 1.67] | 1.36 [1.00 to 1.73] | 1.32 [0.96 to 1.69]
  Week 12: number analyzed (Participants) | 47 | 53 | 41
  Week 12 | 1.28 [0.93 to 1.63] | 1.40 [1.07 to 1.74] | 1.21 [0.83 to 1.59]

13. Secondary Outcome: LS Mean PGI-I of Disability Score at Weeks 4, 8 and 12
Description: An assessment of PGI-I of the participant's disability was conducted by the participant using a 7-point Likert scale ranging from -3= very much worse to +3= very much improved. Higher scores indicate a better outcome. The PGI-I was assessed by the participant answering the following question: "Compared to your disability prior to the study treatment initiation, your disability while performing physical activities (example, standing, walking or running) now is: +3=very much improved; +2=much improved; +1=minimally improved; 0=no change; -1=minimally worse; -2=much worse; -3=very much worse".
Time Frame: Weeks 4, 8 and 12 in the double-blind treatment period
Population: as for outcome 12
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Dysport 300 U | Dysport 500 U
Number analyzed (Participants) | 51 | 53 | 46
units on a scale
  Week 4: number analyzed (Participants) | 51 | 49 | 42
  Week 4 | 1.15 [0.83 to 1.47] | 1.16 [0.83 to 1.48] | 1.31 [0.95 to 1.66]
  Week 8: number analyzed (Participants) | 45 | 47 | 46
  Week 8 | 1.19 [0.85 to 1.53] | 1.23 [0.88 to 1.57] | 1.41 [1.06 to 1.75]
  Week 12: number analyzed (Participants) | 47 | 53 | 41
  Week 12 | 1.15 [0.81 to 1.48] | 1.21 [0.89 to 1.52] | 1.28 [0.92 to 1.64]

14. Secondary Outcome: Mean Change From Baseline in 36-Item Short Form Health Survey (SF-36) Score at Weeks 8 and 12
Description: The SF-36 is a 36-item questionnaire which measures the extent to which physical health impacts an individual's functional ability and perceived wellbeing in mental, social, and physical aspects of life. The SF-36 has 8 subscales: physical function, role physical, bodily pain, global health, vitality, social function, role emotional and mental health. Each scale ranges from 0-100, where 0= lowest level of health and 100= highest level of health. Scores on these subscales can be aggregated into the physical component summary (physical function, role physical, bodily pain and global health) and mental component summary (mental health, vitality, social function and role emotional). Physical component summary score ranges from 0.65 to 80.73 and mental component summary score ranges from -8.81 to 81.65, where low score indicates lowest level of health and high score indicates highest level of health. Positive change from Baseline indicates an improvement in quality of life.
Time Frame: Baseline and Weeks 8 and 12 in the double-blind treatment period
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Dysport 300 U | Dysport 500 U
Number analyzed (Participants) | 58 | 59 | 53
units on a scale
  Week 8: SF-36 - Physical component summary score | 3.08 (7.815) | 3.19 (6.013) | 3.30 (7.127)
  Week 12: SF-36 - Physical component summary score: number analyzed (Participants) | 56 | 58 | 53
  Week 12: SF-36 - Physical component summary score | 3.19 (7.776) | 5.04 (7.430) | 2.51 (7.133)
  Week 8: SF-36 - Mental component summary score | -0.66 (7.299) | -0.30 (6.419) | -0.84 (6.022)
  Week 12: SF-36 - Mental component summary score: number analyzed (Participants) | 56 | 58 | 53
  Week 12: SF-36 - Mental component summary score | -0.43 (5.587) | -0.28 (7.821) | -0.22 (6.970)

ADVERSE EVENTS:
Time Frame: From first administration of study drug (Cycle 1 Day 1) up to end of the study, approximately 36 weeks.
Description: The safety population included all participants who received at least one dose of study drug administration (including only partial administration).
Groups:
- Double-Blind Treatment Period (Cycle 1): Placebo: On Cycle 1 Day 1 in the double-blind treatment period, participants received a single dose of placebo (matching with Dysport) intramuscular injection distributed between 4 injection points in the 4 targeted muscles of the study foot.
  The 4 targeted muscles of the study foot were the oblique head of the adductor hallucis muscle, the transverse head of the adductor hallucis muscle, the flexor hallucis brevis muscle and the extensor hallucis brevis muscle.
- Double-Blind Treatment Period (Cycle 1): Dysport 300 U: On Cycle 1 Day 1 in the double-blind treatment period, participants received a single dose of Dysport 300 U intramuscular injection distributed between 4 injection points (75 U each) in the 4 targeted muscles of the study foot.
  The 4 targeted muscles of the study foot were the oblique head of the adductor hallucis muscle, the transverse head of the adductor hallucis muscle, the flexor hallucis brevis muscle and the extensor hallucis brevis muscle.
- Double-Blind Treatment Period (Cycle 1): Dysport 500 U: On Cycle 1 Day 1 in the double-blind treatment period, participants received a single dose of Dysport 500 U intramuscular injection distributed between 4 injection points (125 U each) in the 4 targeted muscles of the study foot.
  The 4 targeted muscles of the study foot were the oblique head of the adductor hallucis muscle, the transverse head of the adductor hallucis muscle, the flexor hallucis brevis muscle and the extensor hallucis brevis muscle.
- Open-Label Treatment Period (Cycle 2): Dysport 300 U: On Cycle 2 Day 1 in the open-label treatment period, all participants who met retreatment criteria received a single dose of Dysport 300 U intramuscular injection distributed between 4 injection points (75 U each) in the 4 targeted muscles of the study foot.
  The 4 targeted muscles of the study foot were the oblique head of the adductor hallucis muscle, the transverse head of the adductor hallucis muscle, the flexor hallucis brevis muscle and the extensor hallucis brevis muscle.
- Open-Label Treatment Period (Cycle 3): Dysport 300 U: On Cycle 3 Day 1 in the open-label treatment period, all participants who met retreatment criteria received a single dose of Dysport 300 U intramuscular injection distributed between 4 injection points (75 U each) in the 4 targeted muscles of the study foot.
  The 4 targeted muscles of the study foot were the oblique head of the adductor hallucis muscle, the transverse head of the adductor hallucis muscle, the flexor hallucis brevis muscle and the extensor hallucis brevis muscle.
- Open-Label Treatment Period (Cycle 3): Dysport 500 U: On Cycle 3 Day 1 in the open-label treatment period, all participants who met retreatment criteria received a single dose of Dysport 500 U intramuscular injection distributed between 4 injection points (125 U each) in the 4 targeted muscles of the study foot.
  The 4 targeted muscles of the study foot were the oblique head of the adductor hallucis muscle, the transverse head of the adductor hallucis muscle, the flexor hallucis brevis muscle and the extensor hallucis brevis muscle.
Arm/Group | Double-Blind Treatment Period (Cycle 1): Placebo | Double-Blind Treatment Period (Cycle 1): Dysport 300 U | Double-Blind Treatment Period (Cycle 1): Dysport 500 U | Open-Label Treatment Period (Cycle 2): Dysport 300 U | Open-Label Treatment Period (Cycle 3): Dysport 300 U | Open-Label Treatment Period (Cycle 3): Dysport 500 U
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/63 | 0/56 | 0/146 | 0/8 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/63 | 1/56 | 1/146 | 0/8 | 1/56
Other Adverse Events (participants affected / at risk) | 6/61 | 9/63 | 6/56 | 11/146 | 0/8 | 4/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-Blind Treatment Period (Cycle 1): Placebo (N=61) | Double-Blind Treatment Period (Cycle 1): Dysport 300 U (N=63) | Double-Blind Treatment Period (Cycle 1): Dysport 500 U (N=56) | Open-Label Treatment Period (Cycle 2): Dysport 300 U (N=146) | Open-Label Treatment Period (Cycle 3): Dysport 300 U (N=8) | Open-Label Treatment Period (Cycle 3): Dysport 500 U (N=56)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-Blind Treatment Period (Cycle 1): Placebo (N=61) | Double-Blind Treatment Period (Cycle 1): Dysport 300 U (N=63) | Double-Blind Treatment Period (Cycle 1): Dysport 500 U (N=56) | Open-Label Treatment Period (Cycle 2): Dysport 300 U (N=146) | Open-Label Treatment Period (Cycle 3): Dysport 300 U (N=8) | Open-Label Treatment Period (Cycle 3): Dysport 500 U (N=56)
Injection site pain (General disorders) | 1 (1) | 2 (2) | 3 (3) | 3 (4) | 0 (0) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (3) | 3 (5) | 6 (6) | 0 (0) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (5) | 1 (1) | 3 (3) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Based on the results of the primary analysis the sponsor terminated the study early due to lack of efficacy of the tested doses at the primary endpoint. The decision by the sponsor to terminate the study early was not related to any safety or tolerability concerns with Dysport.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-07-03): https://cdn.clinicaltrials.gov/large-docs/98/NCT03569098/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-20): https://cdn.clinicaltrials.gov/large-docs/98/NCT03569098/SAP_001.pdf